CLINICAL TRIAL: NCT01996878
Title: Association Analysis of Single Nucleotide Polymorphisms and the Incidence of Parkinson's Disease in a Hospital-based Case-control Study in Taiwan
Brief Title: Genetic Polymorphism and Parkinson's Disease in Taiwanese
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Shey-Lin Wu, Superintedent, Changhua Christian Hospital
Other Study IDs: CCH060105
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Genetic Polymorphism
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collect 10 mL peripheric blood for DNA extraction

GROUPS / COHORTS (2):
- Case (Parkinson's disease patients): Clinical diagnosis of Parkinson's disease (cases are diagnosed by the presence of at least three of the five following primary signs: rest tremor, bradykinesia, rigidity, impaired postural refluxes, and the presence of a sustained L-dopa response.)
- Control (Healthy volunteers): Healthy volunteers without Parkinson's disease

SUMMARY:
To observe and analyze the correlation between Single Nucleotide polymorphisms (SNPs) and the incidence of Parkinson's disease in Taiwanese.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease (case subjects are diagnosed by the presence of at least three of the five following primary signs: rest tremor, bradykinesia, rigidity, impaired postural refluxes, and the presence of a sustained L-dopa response.)
* Healthy volunteers without Parkinson's disease

Exclusion Criteria:

* Cases showing atypical features, including multiple system atrophy and progressive supranuclear gaze palsy, or secondary causes of Parkinsonism, such as neuroleptic drugs, infection, tumor, previous cerebrovascular accident and known toxins

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Taiwanese
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
single nucleotide polymorphisms in certain candidate genes | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shey-Lin Wu, M.D., Principal Investigator — Chang Hua Christian Hospital
Locations (1):
- Department of Neurology, Chang-Hua Christian Hospital, Chang-hua, Taiwan